CLINICAL TRIAL: NCT06015087
Title: Fasting Diet and Chemotherapy Toxicity
Brief Title: Evaluation of the Influence of Short Term Fasting Diet on Chemotherapy-induced Toxicities in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Odysseas Androutsos, Associate Professor of Clinical Nutrition and Dietetics, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Fasting diet
Record Dates: First submitted 2023-07-25; First posted 2023-08-29 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Fasting, Diet, Chemotherapy, Toxicity
Keywords: fasting diet, breast cancer, chemotherapy toxicity, Mediterranean Diet
MeSH Terms: conditions — Fasting; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: fasting diet
- Control group (No Intervention)

INTERVENTIONS:
Other: fasting diet — A total of 50 patients with breast cancer will be randomly devided in intervention and control group. Intervention group will follow a 60 hours fasting diet (36h prior and 24h after chemotherapy infusion), low in calories, mainly plant based, and the Mediterranean Diet in the meantime between chemotherapy cycles. Control group will receive only standard of care. Nutritional counseling and dietary records will be performed by registered dietitian. Adherence to the Mediterranean Diet will be estimated with MedDietScore. Grade of toxicity will be estimated by using the National Cancer Institute Common Terminology Criteria for Adverse Events. All participants will be encourange to continue usual physical activity.
  Arms: Intervention group

SUMMARY:
This is a clinical trial aiming to assess the effect of fasting diet on chemotherapy - induced toxicities in breast cancer patients. The study will have an intevention group and a control group. The intervention group will follow a fasting diet of 60 hours (36h prior chemotherapy and 24h after the end of chemotherary), while the control group will follow regular (standard) diet. At the meantime of the chemotherapy cycles, the intervention group will be recommended to follow the Mediterranean diet.

The main questions this study is aiming to answer is whether short term fasting diet influences chemotherary - induced toxicities and if it is easy to be implemented.

DETAILED DESCRIPTION:
This is a clinical trial aiming to assess the effect of fasting diet on chemotherapy - induced toxicities in breast cancer patients. The study will have an intevention group and a control group. The intervention group will follow a fasting diet for 60 hours (36h prior chemotherapy and 24h after the end of chemotherapy), while the control group will follow regular diet. At the meantime of the chemotherapy cycles, the intervention group will be recommended to follow the Mediterranean diet. The patients will be randomized in the two groups. A total of 50 patients is required. Biochemical data, anthropometric measures and grading of toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events, nutritional habits, adherence to the Mediterranean diet (implementation of MedDietScore) will be assessed prior, during and after the intervention, in both groups. Nutritional counseling will be performed by Registered Dietitian, and telephone interviews will be used to record adherence to fasting diet and Mediterranean diet.

The main questions this study is aiming to answer is whether short term fasting diet influences chemotherary - induced toxicities and if it is easy to be implemented.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients with first diagnosis of breast cancer
* no distinct metastasis
* patients will receive at least 4 cycles of adjuvant or neo-adjuvant chemotherapy

Exclusion Criteria:

* BMI<19kg/m2
* unintentional weight loss of >3 or >5 kg the last 3 or 6 months respectively
* medical history of anorexia nervosa, boulimia or any other eating disorders
* renal failure (creatinine >2mg/dl)
* diabetes mellitus (type I or Insulin dependent type II)
* serious psychiatric disease
* serious cardiovascular disease
* mobility limitations
* being participant in any other study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the influence of short term fasting diet on the incidence of treatment-emergent adverse events [safety and tolerability]) caused by chemotherapy | The patients with receive 4-8 cycles of chemotherapy,each cycle is repeated every 21 days. At the end of each cycle and prior next cycle the incidence of treatment - emergent adverse events (safety and tolerability) will be accessed.
  Grade of toxicity will be accessed after each chempotherapy, using the National Cancer Institute Common Terminology Criteria for Adverse Events and eorct. Data will be collected and comparison between the two groups will be performed after each chemotherapy cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition-Dietetics, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided